CLINICAL TRIAL: NCT02599870
Title: Prospective Randomized Clinical Study to Evaluate the Clinical Impact of Pharmacogenetics-Guided Treatment for Patients Undergoing Elective Spinal Surgical Procedures
Brief Title: Clinical Study to Evaluate Clinical Impact of PGx-Guided Treatment for Patients Undergoing Elective Spinal Surgical Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: AltheaDx (Industry)
Collaborators: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CLP-0007
Record Dates: First submitted 2015-10-23; First posted 2015-11-09 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Acute Pain; Surgery
Keywords: PGx; pharmacogenetic testing; IDgenetix; Pain Management; AltheaDx; Post-Operative Pain Management
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroIDgenetix Test Panel Intervention (Experimental): The medical provider for the NeuroIDgenetix-guided group will make post-operative pain management recommendations based on test results. Patient outcomes, length of hospital stay and number of medical visits will be measured throughout the study.
  Interventions: Genetic: NeuroIDgenetix Test Panel
- Control (No Intervention): The medical provider for the control group will not receive the NeuroIDgenetix Test Panel results and will make post-operative pain management recommendations based as usual. Patient outcomes, length of hospital stay and number of medical visits will be measured throughout the study.

INTERVENTIONS:
Genetic: NeuroIDgenetix Test Panel — The NeuroIDgenetix Test Panel is used to make recommendations on post-operative pain medication therapy that may be impacted by the genetic background of the patient.
  Other Names: IDgenetix Neuro Test; PGx Testing
  Arms: NeuroIDgenetix Test Panel Intervention

SUMMARY:
The purpose of this study is to evaluate the effect of pharmacogenetic (PGx) guided treatment when implemented into the pre-operative process for patients undergoing an elective spinal surgical procedure and requiring post-operative acute pain management, as compared to a group of subjects with the same attributes without the guidance of PGx testing for their post-surgery pain management. This study will also evaluate whether PGx testing can reduce narcotic consumption, opioid-related adverse effects, time to mobilization, medical visits and costs.

DETAILED DESCRIPTION:
The incidence of opioid related adverse drug events can reach as high as 50% in surgical patients and poor pain management is a significant risk factor for early readmission. In addition, the rate of non- response to certain analgesics is double in patients who are poor metabolizers as demonstrated by mutations in both CPY26d alleles. Finally, there is a growing body of literature that ineffective acute pain management contributes significantly to the risk of chronic pain syndromes. Genetics and drug interactions can alter both the pharmacokinetics and pharmacodynamics of a multitude of drug compounds and in turn influence both the safety and efficacy of selected therapeutic regimens.

Pharmacogenetic-guided therapy selection can enhance patient response by facilitating the selection of the most appropriate medication at the most effective dose in the shortest possible time.

In this prospective, randomized, single-blind study, the investigators will evaluate the clinical impact of pharmacogenetics-guided treatment on the duration of the post-surgical hospital stay and on patient well-being as determined by post-op pain assessments. Additionally, the impact of PGx-guided treatment on narcotic consumption, number of adverse events, re-admission rates and costs will be evaluated during the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over the age of 18;
* Patients undergoing an elective spine surgical procedures
* Willing and able to comply with study procedures
* Able to provide written informed consent
* Surgery timing - scheduled to occur after PGx testing and IDgenetix test report review (at least 4 days after Pre-Op visit)

Exclusion Criteria:

* Unwilling or unable to provide written informed consent and to comply with study procedures
* Any subject for whom providing a buccal swab sample would be contraindicated or not possible
* Subject with a history of chronic renal dysfunction, Chronic Kidney Disease (Stage 4 or 5)
* abnormal hepatic function within the last 2 years (INR >1.2 not attributable to anticoagulant medications, AST/aspartate aminotransferase or ALT/alanine aminotransferase >1.5x normal, or suspected cirrhosis)
* a history of malabsorption (short gut syndrome)
* any gastric or small bowel surgery less than 3 months prior to study enrollment
* Patients with a significant unstable medical condition or life threatening disease
* History of prior pharmacogenetic testing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Comparison of length of post-surgical hospital stay between the two treatment arms. | From date of surgery until hospital discharge, assessed up to 3 months
  Duration of the post-surgical hospital stay
Comparison of patient well being between the two treatment arms as measured by pain scores | 3 months
  Comparison of patient well being between the two treatment arms as measured by pain scores.
Comparison of patient well being between the two treatment arms as measured by disability scores | 3 months
  Comparison of patient well being between the two treatment arms as measured by disability scores.

SECONDARY OUTCOMES:
Comparison of post-operative narcotic consumption between the two treatment arms | 3 months
  Comparison of post-operative narcotic consumption between the two treatment arms
Comparison of opioid-related adverse effects between the two treatment arms | 3 months
  Comparison of opioid-related adverse effects between the two treatment arms
Comparison of time to mobilization between the two treatment arms | 3 months
  Comparison of time to mobilization between the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Wale Sulaiman, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States